CLINICAL TRIAL: NCT06407765
Title: Effects of Dual Task Training With and Without Backward Walking on Balance, Activity and Participation in Children With Cerebral Palsy
Brief Title: Effects of Dual Task Training on Balance, Activity and Participation in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0732
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Dual task training; Backward Walking; Activity; Balance
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: It will be a Randomized control trail. Convenient random sampling is used to collect the sample. The population under study is Cerebral palsy children. The study sample group are between the age of 6 to 12. The group is randomly divided into two groups; Control and experimental group. The control group will receive Dual task training. The experimental group will receive both dual task training and backward walking. The patients will be assesed at the start and then after 4 weeks of treatment.
Who Masked: Participant
Masking Description: Both group will receive separate treatment and effort will be put to mask the both groups about treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Task Training (Active Comparator): This group will receive Dual task training
  Interventions: Other: Dual task training
- Dual task training with Backward walking (Experimental): This group will receive both Dual task training with Backward walking
  Interventions: Other: Dual task training with backward walking

INTERVENTIONS:
Other: Dual task training — Dual task training incorporates both cognitive and motor tasks. Tasks like walking and asking the patient to point towards objects, collect start from the objects hanging above the patient and asking the patient to name the objects shown to him/her. This treatment will be given for 4 weeks, 4 times a week for 40 minutes. Each task is done for 7 minutes with a 3 minutes break in between.
  Arms: Dual Task Training
Other: Dual task training with backward walking — This group will get both dual task training and backward walking. For dual task training same protocol as active comparator is followed. For backward walking; the patient is firstly asked to walk backward with complete physiotherapist assistance. Secondly, the patient is asked to walk for 15 m through the treatment room's hallway while holding a safety bar with the hand on the unaffected side. Third, without using a safety bar, the participants were urged to walk freely. Lastly, the participants tried to walk backwards at a reasonable pace while progressively increasing their distance travelled and speed. This treatment will be given for 4 weeks, 4 times a week for 40 minutes. Each task is done for 7 minutes with a 3 minutes break in between.
  Arms: Dual task training with Backward walking

SUMMARY:
Cerebral palsy is a non progressive neurodevelopmental disorder that usually effects the muscles of the patients effecting its tone, strength and eventually ability to move. Dual tasking training incorporates more than one task at a time, it can b either physical task with movement or mental tasks. Backward walking is used to challenge the proprioception.

The study is a randomized controlled trial to assess the effects of Dual task training with and without Backward walking on balance, activity and participations on children with cerebral palsy. Study will be conducted in PSRD and Rehab care. Sample will be recruited randomly and then divided into two groups control and experimental group. Control group will receive dual task training and experimental group will receive both dual task training and backward walking. This treatment would continue for 4 weeks. Patient will be assessed both at the start and end of 4 weeks. The outcome tools for assessment of balance, activity and participation will be following: Pediatric Berg Balance Scale, Time up and Go test and Participation of daily life PODCI Questionnaire. Ethical consideration will be followed and informed consent will be taken from legal guardians.

DETAILED DESCRIPTION:
The randomized control trail includes two groups; Control and experimental group. Control group will receive Dual task training. Dual task training incorporates cognitive and motor task. motor task like waking on balance beam is combined with visual memory tasks like pointing towards an object the therapists asks, ask the patient to collect the hanging stars while different shapes are hanging above him, name the object in the picture shown to patient. This treatment will continue for 4 weeks, 4 times a week for 40 minutes.

Experimental group will receive both Dual task training and Backward walking. with the activities mentioned above patient will be asked to walk backward with any obstacle firstly with complete physiotherapist assistance and then gradually with less assistance. Secondly patients will be asked to cover a distance of 15 m through the treatment room's hallway while holding a safety bar with the hand on the unaffected side. Third, without using a safety bar, the participants were urged to walk freely. Lastly, the participants tried to walk backwards at a reasonable pace while progressively increasing their distance travelled and speed. the duration of the treatment will be the same. The patients will be assessed first at the start of treatment and then at the end of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy who have already received a diagnosis
* Children with GMFCS Level I-II
* Children between the ages of 6 and 12

Exclusion Criteria:

* Being unable to complete the cognitive task, which involves counting back one after each number between 0 and 100
* Posing a behavioral issue that makes it challenging to engage in the study
* Being unable to walk independently
* Children with concomitant cardiac conditions
* Any musculoskeletal surgery performed during the previous six months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale | 4 weeks
  A version of Berg's Balance Scale, the Pediatrics Balance Scale (PBS) was created as a balancing assessment for school-age children with mild to moderate motor deficits. There is a 0.998 intra-class correlation value (ICC).
Time up and go test | 4 weeks
  In clinical practice, the "timed up and go" (TUG) test is a brief assessment tool used to evaluate adults' functional mobility. The TUG test has a high level of dependability in children as well, with an ICC of 0.99 both within a session and between tests.
Participation of Daily Life PODCI Questionnaire | 4 weeks
  The PODCI is a parent-reported outcome measure that evaluates children's expectations of healthcare interventions as well as their mobility, physical function, comfort, and happiness. When assessing quality of life issues and walking function in children with cerebral palsy, the PODCI shows good validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Aqsa Butt, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher-Pipher S Pt Dpt, Kenyon LK Pt Dpt PhD Pcs, Westman M Pt Dpt. Improving balance, mobility, and dual-task performance in an adolescent with cerebral palsy: A case report. Physiother Theory Pract. 2017 Jul;33(7):586-595. doi: 10.1080/09593985.2017.1323359. Epub 2017 May 16. PMID 28509631